CLINICAL TRIAL: NCT01114347
Title: Prevention of Nosocomial Escherichia Coli Infections After Placement of an Indwelling Catheter During Pelvic Surgery: a Randomized, Prospective, Double Blind Study for the Evaluation of Cranberry (Vaccinium Macrocarpon) Gel Capsules
Brief Title: Prevention of Nosocomial E. Coli Infections After Placement of an Indwelling Catheter During Pelvic Surgery: an Evaluation of Cranberry Gel Capsules
Acronym: NosoPink
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AOI/2009/VL-01; 2009-A01317-50 (Other: ANSM)
Record Dates: First submitted 2010-04-30; First posted 2010-05-03 (Estimated); Last update posted 2025-11-17 (Actual); Status verified 2015-03

CONDITIONS: Cross Infection; Bacteriuria
MeSH Terms: conditions — Cross Infection; Bacteriuria

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cranberry (Experimental): Patients randomized to this arm will recieve one gel capsule containing cranberry PAC (36 mg of type A pro anthocyandines: Urell, Pharmatoka) per day starting at the day of the pelvic surgery (j0) until day 10 postop (j10). The gel capsule in taken orally in the morning with a large glass of water.
  Interventions: Dietary Supplement: cranberry type A pro anthocyandines
- Placebo (Placebo Comparator): The patients randomized to this arm will recieve one placebo gel capsule per day starting on the day of the pelvic surgery (j0) until the 10th day post-op (j10). The gel capsule is taken orally in the morning with a large glass of water. The placebo contains lactose and is conditioned in a manner to be identical in caliber and color with the experimental treatment gel capsules.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: cranberry type A pro anthocyandines — One gel capsule containing cranberry PAC (36 mg of type A pro anthocyandines: Urell, Pharmatoka) per day starting at the day of the pelvic surgery (j0) until day 10 postop (j10). The gel capsule in taken orally in the morning with a large glass of water
  Arms: Cranberry
Dietary Supplement: Placebo — One placebo gel capsule per day starting on the day of the pelvic surgery (j0) until the 10th day post-op (j10). The gel capsule is taken orally in the morning with a large glass of water. The placebo contains lactose and is conditioned in a manner to be identical in caliber and color with the experimental treatment gel capsules.
  Arms: Placebo

SUMMARY:
Indwelling urinary catheters are a primary site for nosocomial infections. The purpose of this study is to evaluate the anti-adhesive properties of Cranberry type A pro anthocyanidine gel capsules in the prevention Escherichia coli infections on indwelling urinary catheters placed in patients following pelvic surgery. The investigators primary working hypothesis is that cranberry treatment decreases E. coli colonization on indwelling urinary catheters, thus preventing nosocomial urinary infections following pelvic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patient is cared for by the department of the Gynecology at the Nîmes Unversity Hospital
* The patient is programmed for surgery with placement an indwelling catheter for 48 hours with a sterile urinary cytobacteriologic exam at inclusion

Exclusion Criteria:

* the urinary cytobacteriologic exam at inclusion is positive
* the patient is taking antivitamin K
* the patient is taking antibiotics
* history of urolithiasis
* the patient refuses to participate
* the patient is pregnant or nursing
* the patient is not associated with a social security system (no insurance)
* the patient is under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2010-08; Primary Completion 2014-03-22 (Actual); Study Completion 2014-03-22 (Actual)

PRIMARY OUTCOMES:
Presence/absence of Asymptomatic bacteriuria | 15 days post-op
  Presence/absence of greater than 10^5 unit forming E. coli colonies per ml of urine with absence of functional urinary infection symptoms (mictional burning, pollakiuria, dysuria, urgency, suprapubic heaviness)

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Letouzey, MD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (1):
- CHU de Nîmes - Hôpital Universitaire Carémeau, Nîmes, France

REFERENCES:
- [Result] Letouzey V, Ulrich D, Demattei C, Alonso S, Huberlant S, Lavigne JP, de Tayrac R. Cranberry capsules to prevent nosocomial urinary tract bacteriuria after pelvic surgery: a randomised controlled trial. BJOG. 2017 May;124(6):912-917. doi: 10.1111/1471-0528.14524. Epub 2017 Feb 10. PMID 28186383
- [Derived] Williams G, Stothart CI, Hahn D, Stephens JH, Craig JC, Hodson EM. Cranberries for preventing urinary tract infections. Cochrane Database Syst Rev. 2023 Nov 10;11(11):CD001321. doi: 10.1002/14651858.CD001321.pub7. PMID 37947276
- [Derived] Williams G, Hahn D, Stephens JH, Craig JC, Hodson EM. Cranberries for preventing urinary tract infections. Cochrane Database Syst Rev. 2023 Apr 17;4(4):CD001321. doi: 10.1002/14651858.CD001321.pub6. PMID 37068952